CLINICAL TRIAL: NCT04813315
Title: Effects of Kendall Exercise Versus Gong's Mobilization on Pain, Range of Motion, Function and Strength in Text Neck Syndrome. A Pilot Study
Brief Title: Effects of Kendall Exercise Versus Gong's Mobilization in Text Neck Syndrome. A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/0105
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Neck Pain
Keywords: neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kendall exercise (Experimental): Experimental group 1 got this intervention containing Kendall exercise for 15-20 mins, followed by conventional physiotherapy treatment (hot pack).Participants were treated 3 times per week for 4 weeks. Pre and Post treatment readings were taken in 1st session and 4th week respectively. Assessment was done via Numeric pain rating scale, neck disability index, universal goniometer and modified sphygmomanometer test.
  Interventions: Other: Kendall exercise
- Gong's mobilization (Experimental): Experimental group 1 got this intervention containing Gong's mobilization for 15-20 mins, followed by conventional physiotherapy treatment (hot pack).Participants were treated 3 times per week for 4 weeks. Pre and Post treatment readings were taken in 1st session and 4th week respectively. Assessment was done via Numeric pain rating scale, neck disability index, universal goniometer and modified sphygmomanometer test.
  Interventions: Other: Gong's mobilization

INTERVENTIONS:
Other: Kendall exercise — consist of stretch of pectoralis major and neck extensor strengthening of deep neck flexors and scapular retractor
  Arms: Kendall exercise
Other: Gong's mobilization — it is combination of glide along the facet joint and concurrent movement of cervical spine
  Arms: Gong's mobilization

SUMMARY:
This project was a pilot randomized trial conducted to compare the effects of Kendall exercise and Gong's mobilization on pain, range of motion, function and strength in text neck syndrome so that we can have best treatment option for patients with neck pain

DETAILED DESCRIPTION:
Non Probability Convenient sampling was done. Patients following eligibility criteria from Fatima hospital Sargodha were considered. Sample size was calculated 12.

Participants were randomly allocated in two groups equally via convenient sampling method. Baseline assessment was done initially. Group A was given Kendall exercise and Group B was given Gong's mobilization along with conventional physiotherapy treatment (hot pack). Duration of research was almost 6 months. Participants were treated 3 times a week for 4 weeks. Pre and Post treatment readings were taken in 1st session and 4th week period respectively.

Assessment was done via Numeric pain rating scale (NPRS),Neck Disability index (NDI), Universal goniometer and Modified sphygmomanometer test. All participants were provided written informed consent prior to commencement of the procedures. They were free to quit the treatment at any stage of research. Data was analyzed by using SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

* Young adults
* more than one year using a smartphone
* Using smart phone for more than 2 hours a day
* Craniovertebral angle(CVA)less than 53°
* Score of more than 3 on NPRS and more than 10 on NDI

Exclusion Criteria:

* Spinal infection or inflammatory disorder
* Neck surgery or trauma
* Torticollis, scoliosis
* Malignancy, pregnancy
* Diagnosed cases of disc prolapse, stenosis, herniation, spondylolisthesis and osteoporosis
* Current use of any medication or physical therapy treatment.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4th week
  Numeric pain rating scale range from 0-10, 0 means no pain- 10 means severe pain First checked at baseline and than 4th week
Range of Motion | 4th week
  All ranges of neck: 80° to 90° of flexion, 70° of extension, 20° to 45° of lateral flexion, and up to 90° of rotation to both sides. All ranges other than the written will be considered abnormal.
  First checked at baseline and than 4th week
Neck Disability Index | 4th week
  Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. o means no pain 5 means maximum pain Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50.0 means no disability, 50 means full limitation.A higher score indicates more patient-rated disability.
  First checked at baseline and than 4th week
Modified Sphygmomanometer test | 4th week
  It is used to measure strength of muscles. change in 2mm cause minimal detectable change.
  First checked at baseline and than 4th week

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah IU, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim KH, Kim SG, Hwangbo G. The effects of horse-riding simulator exercise and Kendall exercise on the forward head posture. J Phys Ther Sci. 2015 Apr;27(4):1125-7. doi: 10.1589/jpts.27.1125. Epub 2015 Apr 30. PMID 25995571
- [Background] Neupane S, Ali UI, Mathew A. Text neck syndrome-systematic review. Imperial Journal of Interdisciplinary Research. 2017;3(7):141-8.
- [Background] Gong W. The effects of cervical joint manipulation, based on passive motion analysis, on cervical lordosis, forward head posture, and cervical ROM in university students with abnormal posture of the cervical spine. J Phys Ther Sci. 2015 May;27(5):1609-11. doi: 10.1589/jpts.27.1609. Epub 2015 May 26. PMID 26157273